CLINICAL TRIAL: NCT06087887
Title: Association Between Tumor Size and Prognosis in Patients With Small Bowel adenocarcinoma-a SEER-based Study
Status: Completed | Type: Observational
Sponsor: Zhe Fan (Other)
Responsible Party: Sponsor-Investigator, Zhe Fan, docter, The Third Peoples Hospital of Dalian
Organization: The Third Peoples Hospital of Dalian (Other)
Other Study IDs: ThirdPHDalian
Record Dates: First submitted 2023-10-11; First posted 2023-10-18 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Prognosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- tumor size 0-1cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 0-1 cm.
  Interventions: Other: no interventions
- tumor size 1-2 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 1-2 cm.
- tumor size 2-3 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 2-3 cm.
- tumor size 3-4 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 3-4 cm.
- tumor size 4-5 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 4-5 cm.
- tumor size 5-6 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 5-6 cm.
- tumor size 6-7 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 6-7 cm.
- tumor size 7-8 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 7-8 cm.
- tumor size 8-9 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 8-9 cm.
- tumor size 9-10 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of 9-10 cm.
- tumor size >10 cm: No intervention. Select small bowel adenocarcinoma patients with tumor size of >10 cm.

INTERVENTIONS:
Other: no interventions — no interventions
  Groups: tumor size 0-1cm

SUMMARY:
The goal of this observational study is to learn about in small bowel adenocarcinoma patients. The main question it aims to answer is the association between tumor size and prognosis in patients with small bowel adenocarcinoma. Participants will be compared for the relationship between tumor size and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. pathology confirmed as SBA;
2. received surgery and complete postoperative follow-up data;
3. histology type code 8140-8380.

Exclusion Criteria:

Cases with unknown tumor location, size, TNM staging, race, and degree of differentiation were excluded. Finally, 8,163 eligible patients were included in the analysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data of Small Bowel adenocarcinoma patients from 2004 to 2019 was collected from the SEER database using the SEER*Stat software (version 8.4.0.1).
Sampling Method: Non-Probability Sample
Enrollment: 8163 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Association Between Tumor Size and Prognosis in Patients With Small Bowel adenocarcinoma-a SEER-based Study | 2024.9.1
  We will study the relationship between tumor size and prognosis in small bowel adenocarcinoma patients in the SEER database

CONTACTS AND LOCATIONS:
Locations (1):
- Dalian Third People's Hospital Affiliated to Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes